CLINICAL TRIAL: NCT03803007
Title: Randomized, Double Blind, Multi Center, Multinational, Placebo Controlled, Single Parallel Escalating Dose Safety and Efficacy Study of ACT017 Used as an Add on Therapy on Top of Standard of Care of Acute Ischemic Stroke
Brief Title: Acute Ischemic Stroke Interventional Study
Acronym: ACTIMIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acticor Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT-CS-002; 2018-002855-13 (EudraCT Number)
Record Dates: First submitted 2018-12-12; First posted 2019-01-14 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Haemorrhages; Thrombolysis; Thrombectomy; Anti-platelet; glenzocimab; ACT017; stroke; GPVI
MeSH Terms: conditions — Ischemic Stroke; Hemorrhage; Stroke

STUDY DESIGN:
Intervention Model Description: The phase Ib of the study with a sequential design has been achieved (5 arms). The second phase IIa is ongoing. The selected dose (1000mg) for this second part will be compared to placebo (2 arms) with a parallel design.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous glenzocimab (ACT017) 1000 mg (Experimental): Intravenous glenzocimab (ACT017) 1000 mg to be added to a tissue plasminogen activator +/- mechanical thrombectomy
  Interventions: Drug: Intravenous ACT017 1000 mg
- Intravenous Placebo (Placebo Comparator): Intravenous Placebo to be added to a tissue plasminogen activator +/- mechanical thrombectomy
  Interventions: Other: Intravenous Placebo

INTERVENTIONS:
Drug: Intravenous ACT017 1000 mg — Add-on therapy to the standard of Care in the treatment of the acute ischemic stroke symptoms
  Other Names: Thrombolysis by rtPA +/- thrombectomy
  Arms: Intravenous glenzocimab (ACT017) 1000 mg
Other: Intravenous Placebo — Add-on therapy to the standard of Care in the treatment of the acute ischemic stroke symptoms
  Other Names: Thrombolysis by rtPA +/- thrombectomy
  Arms: Intravenous Placebo

SUMMARY:
To assess safety of single IV (bolus + infusion) doses of ACT017 in patients with an acute ischemic stroke in addition to best emergency standard of care (including fibrinolysis by rtPA with or without added thrombectomy), with a specific focus on hemorrhage, whether clinically symptomatic (NIHSS score + 4 points or death, without other explanation), or seen (excluding other diagnoses) on 24-hour (hr) CT scan, serious adverse events (SAEs), suspected unexpected serious adverse reactions (SUSARs), and medically important events and other safety items including biological and immunological tolerability.

DETAILED DESCRIPTION:
This first in-patient randomized, double blind, multicenter, multinational, placebo-controlled, parallel-dose 2-phase study combines a dose-escalation phase (1b) and a consolidation phase (2a).

Dose Escalation (Phase 1b):

Phase 1b was designed to (I) assess the dose- related safety and potential efficacy of glenzocimab administered as soon as possible and no later than 3 hours after the start of thrombolysis with tPA (itself administered within 4.5 hrs of the onset of acute ischemic stroke symptoms), and (II) identify the recommended phase 2 dose (RP2D).

During this phase, patients were unevenly randomized between groups, to obtain a total of 60 patients, 12 at each dose level. At the starting level, 8 patients received either glenzocimab at the lowest pharmacologically active dose of 125 mg (n=4) or the matching placebo(n=4). After real-time review by the DSMB of clinical safety and a CT scan (and where available MRI) and giving a favorable opinion, the next patients were randomized in the second cohort (n=8) with 4 patients under a higher dose of 250 mg, 2 patients remaining at the initial starting dose (125 mg), and 2 patients under placebo. Following the same process, and after favorable opinion from the DSMB, patients were randomized in the third cohort (n=10) and received glenzocimab 500 mg (n=4), randomized versus 250 mg (n=2), 125 mg (n=2) or placebo (n=2). Similarly, the fourth cohort (n=12) randomized patients between ahigher dose of 1000 mg (n=4), versus 500 mg (n=2), 250 mg (n=2), 125 mg (n=2), or placebo (n=2). Once this fourth cohort completed, the DSMB issued a further positive opinion and the fifth cohort (n=22) randomized patients to 1000 mg (n=8), versus 500 mg (n=6), 250 mg (n=4), 125 mg (n=2), or placebo (n=2).

Consolidation Phase with Final Dose (Phase 2a):

After having reviewed patient's safety data included in the first part of the study, the DSMB confirmed that the study can continue with the glenzocimab recommended dose of 1000 mg. During this phase, a group of 100 patients will be treated, 50 with glenzocimab and 50 with matching placebo to complete the group of 160 patients planned to participate in this study.

In addition, patients in each treatment arm will be stratified by type of Standard of Care (SOC) administered:

* Thrombolysis with tPA only;
* Thrombolysis with tPA AND mechanical thrombectomy Each treatment arm will contain 25 patients with one SOC, and 25 with the other SOC. The active glenzocimab dose will be that recommended after the last safety analysis has been performed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients ≥ 18 years (i.e., at least 18 years old at time of randomization). Extreme caution should be exercised in patients over 80 years of age with regards their general health, neurological status and any concomitant diseases and treatments that are likely to be more common;
2. Patients who have given written consent, legal representative consent or emergency consent (including e-consent) in accordance with local legal and IECs/IRBs requirements;
3. Patients presenting with an acute disabling ischemic stroke in either the anterior or posterior circulation.The time of onset is known or if unknown, the last time the patient was seen well, was at most 4.5 hrs before confirmation of the diagnosis enabling the initiation of alteplase administration within this time-frame;
4. Patients presenting at least a NIHSS ≥ 6 prior to thrombolysis with tPA;
5. Patients eligible for, or administered thrombolysis treatment with tPA;
6. Patients who can undergo mechanical thrombectomy if eligible;
7. Patients affiliated to social security insurance (if applicable, in accordance to local regulations);
8. Effective birth control method should be used for at least the next 2 months by women, and 4 months by men after IMP administration; birth control methods considered to be highly effective include:

   * intrauterine device
   * intrauterine hormone-releasing system
   * bilateral tubal occlusion
   * vasectomized partner
   * sexual abstinence (if applicable in accordance to local regulations)
9. Women of child-bearing potential must undergo a urinary or plasma pregnancy test with negative results;

Exclusion Criteria:

1. Coma, and/or NIHSS >25;
2. Patients < 18 years of age;
3. Prior ischemic stroke within the past 3 months with pre-stroke mRS known to be > 2;
4. Baseline CT-scan evaluation: more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline imaging;
5. Significant mass effect with midline shift;
6. Stroke of hemorrhagic origin;
7. Contra-indications to thrombolysis with tPA:

   1. Patients with known hypersensitivity to the active substance alteplase or to any of its excipients;
   2. Patients with a high risk of hemorrhages:

      * significant bleeding disorder at present or within the past 6 months;
      * known haemorrhagic diathesis (episodes within past 6 months);
      * patients receiving effective oral anticoagulant treatment, e.g. warfarin sodium;
      * manifest or recent severe or dangerous bleeding;
      * known history of or suspected intra-cranial haemorrhage;
      * any history of central nervous system lesion (i.e. trauma, intra-parenchymal neoplasm, unsecured aneurysm, intracranial or spinal surgery, vascular malformation etc..);
      * recent (< 10 days) traumatic external heart massage, obstetrical delivery, or puncture of a non-compressible blood-vessel (e.g. subclavian or jugular vein puncture);
      * bacterial endocarditis, pericarditis;
      * acute pancreatitis;
      * documented ulcerative gastrointestinal disease during the past 3 months, oesophageal varices, arterial-aneurysm, arterial/venous malformations;
      * neoplasm involving an increased risk of bleeding;
      * severe liver disease, including hepatic failure, cirrhosis, portal hypertension (esophageal varices) and active hepatitis;
      * major surgery or significant trauma during the past 3 months;
      * patients receiving anti-coagulants prior to study: the inclusion may however be considered when the dose or time since the last intake of anticoagulant treatment makes residual efficacy unlikely. This should be confirmed by the appropriate tests of anticoagulant activity for the product(s) concerned to show no clinically relevant activity on the coagulation system defined as follows :

        * INR ≤ 1.5 for vitamin K antagonists; .
        * Low Molecular Weight Heparin (LMWH) and Unfractionated Heparin (UFH): aPPT/ACT/KCT ≤ 39 sec or their patient/witness ratio ≤ 1.2 and/or PT ≤ 16 sec (heparin at sub-therapeutic doses (≤ 50 IU/kg) during the mechanical thrombectomy procedure is authorized);
        * Non-Vitamin-K or Direct Oral Anti-Coagulants (NOACs- DOACs) ≤ 50 ng/mL in patients with normal renal function;
      * need for carotid stenting together with a dual anti-platelet treatment (on top of glenzocimab); this can be carried out 24 hrs after the initiation of treatment with glenzocimab;
      * platelets count <100 × 103/μL (<100 000/ mm3)
      * prior hemorrhagic stroke.
   3. Systolic blood pressure ≥ 185 mm Hg despite appropriate acute therapy to lower blood pressure therapy;
   4. Diastolic blood pressure ≥ 110 mm Hg; despite appropriate acute therapy to lower blood pressure therapy;
   5. Glucose >400 mg/dL (>4 g/L) despite treatment;
   6. Glycemia <50 mg/dL (<0,5 g/L);
8. Patients receiving a dual antiplatelet treatment;
9. Cardiopulmonary resuscitation within the past 10 days;
10. Childbirth within the past 10 days,
11. Epileptic seizure at the onset of symptoms;
12. Life expectancy < 3 months
13. Pregnant or breastfeeding;
14. Females of childbearing potential not using effective birth control methods;
15. Known severe (grade 3 and above) renal impairment or Glomerular Filtration Rate < 30 ml/min/1.73 m2 or Serum Creatinine > 2X ULN (1.2 mg/dL for men and 1.0 mg/dL for women) at screening;
16. Known current participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Symptomatic intracranial haemorrhages | 24 hours
  Number of participants experiencing a symptomatic haemorrhage defined by a secondary increase in National Institute Health Stroke Scale score by 4 points or greater, or death
Incidence of non-symptomatic intracranial haemorrhages | 24 hours
  Non-symptomatic haemorrhages are those detected by Computerized Tomography scan

SECONDARY OUTCOMES:
Change from baseline of National Institute Health Stroke Scale score (7 minimum, 42 maximum), brain lesions and vessel recanalization | 24 hours
  Absolute change from baseline of National Institute Health Stroke Scale score, change from baseline on brain lesions as assessed by Computerized Tomography scan or Magnetic Resonance Imaging or Magnetic Resonance Angiography, change from baseline on Recanalization as measured by the modified Thrombolysis In Cerebral Infarction score (0 minimum, 3 maximum) on Magnetic Resonance Angiography
Change from baseline of National Institute Health Stroke Scale score (7 minimum, 42 maximum), brain lesions and vessel recanalization | 24 hours
  Relative (%) change from baseline of National Institute Health Stroke Scale score, change from baseline on brain lesions as assessed by Computerized Tomography scan or Magnetic Resonance Imaging or Magnetic Resonance Angiography, change from baseline on Recanalization as measured by the modified Thrombolysis In Cerebral Infarction score (0 minimum, 3 maximum) on Magnetic Resonance Angiography
Change from baseline of modified Ranking Scale score assessment | Day 90
  modified Ranking Scale score (0 minimum and 6 maximum): number of patients with favorable outcome (score 0-2)
Change from baseline of modified Ranking Scale score assessment | Day 90
  modified Ranking Scale score (0 minimum and 6 maximum): percentage of patients with favorable outcome (score 0-2)
Change from baseline on size of infarct zone | Day 7
  Change from baseline on size of infarct zone assessed by a central Magnetic Resonance Imaging review
Change from baseline on vital signs | 6 hours, 24 hours, Day 7, Day 30 and Day 90
  Change from baseline on systolic and diastolic blood pressure
Change from baseline on vital signs | 6 hours, 24 hours, Day 7, Day 30 and Day 90
  Change from baseline on heart rate
Change from baseline on clinical laboratory assessments | Day 90
  Change from baseline on plasma haemoglobin level
Change from baseline on clinical laboratory assessments | Day 90
  Change from baseline on platelet count
Change from baseline on clinical laboratory assessments | Day 90
  Change from baseline on serum glucose concentration
Change from baseline on clinical laboratory assessments | Day 90
  Change from baseline on serum creatinine concentration
Change from baseline on ElectroCardioGram (ECG) | 24 hours and Day 90
  Change from baseline on 12-lead ElectroCardioGram (ECG)
Evidence of anti-ACT017 antibodies (ADA) | Day 30 and Day 90
  To assess evidence of anti-ACT017 antibodies (ADA) as a possible to ACT017 administration
Pharmacokinetics on ACT017 plasma concentration | 30 minutes, 9 hours and 24 hours
  Change from baseline on ACT017 plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Comenducci, MD, Study Director — Acticor Biotech
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux,, Bordeau, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voors-Pette C, Lebozec K, Dogterom P, Jullien L, Billiald P, Ferlan P, Renaud L, Favre-Bulle O, Avenard G, Machacek M, Pletan Y, Jandrot-Perrus M. Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of ACT017, an Antiplatelet GPVI (Glycoprotein VI) Fab. Arterioscler Thromb Vasc Biol. 2019 May;39(5):956-964. doi: 10.1161/ATVBAHA.118.312314. PMID 31017822
- [Background] Renaud L, Lebozec K, Voors-Pette C, Dogterom P, Billiald P, Jandrot Perrus M, Pletan Y, Machacek M. Population Pharmacokinetic/Pharmacodynamic Modeling of Glenzocimab (ACT017) a Glycoprotein VI Inhibitor of Collagen-Induced Platelet Aggregation. J Clin Pharmacol. 2020 Sep;60(9):1198-1208. doi: 10.1002/jcph.1616. Epub 2020 Jun 4. PMID 32500636
- [Derived] Mazighi M, Kohrmann M, Lemmens R, Lyrer PA, Molina CA, Richard S, Toni D, Pletan Y, Sari A, Meilhoc A, Jandrot-Perrus M, Binay S, Avenard G, Comenducci A, Grouin JM, Grotta JC; ACTIMIS Study Group. Safety and efficacy of platelet glycoprotein VI inhibition in acute ischaemic stroke (ACTIMIS): a randomised, double-blind, placebo-controlled, phase 1b/2a trial. Lancet Neurol. 2024 Feb;23(2):157-167. doi: 10.1016/S1474-4422(23)00427-1. PMID 38267188